CLINICAL TRIAL: NCT07089797
Title: Effect of Nurse-supported Mobile App for Self-help Cognitive Behavioral Therapy for Insomnia in Informal Cancer Caregivers: a Randomized Controlled Trial
Brief Title: Nurse-supported Mobile App for Self-help CBT-I in Informal Cancer Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yangxi Huang, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nurse-supported CBT-I (FULL)
Record Dates: First submitted 2025-07-25; First posted 2025-07-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Insomnia Chronic; Cancer Caregivers
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nurse-Supported Mobile App for Self-Help CBT-I in Cancer Caregivers (Experimental)
  Interventions: Behavioral: Nurse-Supported Mobile App for Self-Help CBT-I
- Sleep hygiene education (Active Comparator)
  Interventions: Behavioral: Sleep hygiene education

INTERVENTIONS:
Behavioral: Nurse-Supported Mobile App for Self-Help CBT-I — The intervention consists of two components: 1) a mobile app (i.e., WeChat mini program) delivered 6-week self-help CBT-I program; and 2) Weekly nurse support session (up to 20 minutes each) across a 6 week intervention period.
  Arms: Nurse-Supported Mobile App for Self-Help CBT-I in Cancer Caregivers
Behavioral: Sleep hygiene education — The participants in the control group will receive only sleep hygiene (one-page handout) via WeChat. Access to the CBT-I WeChat mini program will be offered to these participants after the completion of the 3-month follow-up assessment.
  Arms: Sleep hygiene education

SUMMARY:
This mixed-methods randomized controlled trial investigates whether a nurse-supported mobile app for self-help cognitive behavioral therapy for insomnia (CBT-I) effectively reduces insomnia severity among informal cancer caregivers, compared to sleep hygiene education.<br><br>

The primary research question is:<br> Does nurse-supported mobile app for self-help CBT-I lower insomnia severity among cancer caregivers compared to sleep hygiene education at post-intervention and 3-month follow-up?<br><br>

A total of 208 participants will:<br>

1. Be randomly assigned to one of two groups:<br> (i) the nurse-supported mobile app-based self-help CBT-I group, which involves a 6-week CBT-I program delivered via a WeChat mini program along with weekly nurse support sessions (up to 20 minutes each); or<br> (ii) the sleep hygiene education group.<br>
2. Complete assessments at baseline, post-intervention, and 3-month follow-up to measure changes in insomnia severity (primary outcome). Secondary outcomes include subjective sleep outcomes, psychological well-being, caregiver burden, fatigue, health-related quality of life, and participants' acceptability and satisfaction.<br><br>

As recommended for trials of complex interventions, investigators will conduct a process evaluation in alignment with the Medical Research Council (MRC) guidance. The key functions of the process evaluation include: *(1) implementation, (2) mechanisms of impact, and (3) context.*

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informal caregiver (e.g., family member or a friend) who co-resides with a cancer survivor of any site or stage and provides at least 4 hours of unpaid daily care. If two or more caregivers are available for a cancer survivor, the one providing most of the daily care will be included.
* Able to understand the research procedures, and read and communicate in Chinese
* Able to use WeChat
* Insomnia severity index scores > 7

Exclusion Criteria:

* Another sleep disorder (e.g., obstructive sleep apnea, restless leg syndrome, rapid eye movement behavior disorder), besides insomnia, that is not adequately treated
* Psychotic disorders (e.g., bipolar disorder, schizophrenia); Suicidal ideation with intent and plan OR attempted suicide within the past 2 months
* Currently taking any psychotropic drugs (e.g., antidepressants, anxiolytics, sleep medications)
* Unstable or acute medical condition or condition requiring surgery in the next 6 months; Pregnancy; or Epilepsy
* Currently participating in any other interventional program
* Prior experience with CBT-I
* Night, evening, early morning or rotating shift work
* Currently caring for a cancer patient receiving hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity | Baseline to 18 week
  Insomnia severity will be assessed by Insomnia Severity Index (ISI). The ISI is a well-validated, 7-item scale designed to assess the severity of insomnia retrospectively over the past 2 weeks. Total scores range from 0 to 28, with higher scores indicating more severe insomnia symptoms.

SECONDARY OUTCOMES:
Sleep patterns | Baseline to 18 week
  Sleep patterns (i.e., total sleep time [TST], time in bed [TIB], sleep efficiency [SE], wake after sleep onset [WASO], and sleep onset latency [SOL]) will be assessed using the Consensus Sleep Diary (CSD). The CSD is widely used to assess subjective sleep parameters.
Sleep quality | Baseline to 18 week
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a widely used, 19-item questionnaire designed to measure various aspects of sleep quality over the past month. Scores range from 0 to 21, with higher scores indicating poorer sleep quality.
Caregiver burden | Baseline to 18 week
  The caregiver burden will be evaluated by Zarit Burden Interview-12 (ZBI-12). The ZBI-12 is a widely used, 12-item shortened version of the original ZBI, designed to assess the subjective burden experienced by informal caregivers. Total scores range from 0 to 48, with higher scores indicating a greater level of caregiver burden.
Depressive symptoms | Baseline to 18 week
  Depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a widely used, 9-item questionnaire designed to screen for, diagnose, monitor, and measure the severity of depression. Each item evaluates the frequency of depressive symptoms experienced over the past two weeks. Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Anxiety symptoms | Baseline to 18 week
  Anxiety symptoms will be assessed using the Generalized Anxiety Disorder-7 (GAD-7). This self-administered, 7-item questionnaire was designed as a screening tool and a severity measure for GAD. Each item asks about the frequency of anxiety symptoms over the past two weeks. Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Fatigue | Baseline to 18 week
  Fatigue will be assessed using the Multi-Dimensional Fatigue Inventory (MFI). The MFI is a 20-item self-report questionnaire designed to measure five dimensions of fatigue (i.e., general fatigue, mental fatigue, physical fatigue, reduced activity, and reduced motivation). Total scores range from 20 to 100, with higher scores indicating greater levels of fatigue.
Health-related quality of life | Baseline to 18 week
  Health-related quality of life will be assessed using the five-dimension five-level European Quality of Life scale (EQ-5D-5L). The EQ-5D-5L is a standardized questionnaire designed to evaluate five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L score ranges from -0.39 to 1, with higher scores indicating better quality of life. Additionally, the EQ-5D-5L includes a Visual Analog Scale (VAS) for overall self-rated health status, with scores ranging from 0 to 100, where higher scores represent better health-related quality of life.
Participants' acceptability and satisfaction | Week 6 to week 18
  The participants' perspectives of acceptability and satisfaction will be evaluated using eight adapted items from the Acceptability E-scale. Each item is rated on a 5-point Likert scale, with scores ranging from 1 to 5. The total score ranges from 8 to 40, with higher scores indicating greater acceptability and satisfaction with the intervention.
Adverse events | Baseline to 18 week
  All adverse events reported by the participants will be documented.
Intervention delivery | Six weeks post-randomization
  The delivery of the intervention will be assessed via semi-structured qualitative interviews conducted with trial participants after the intervention. Intervention adherence will also be assessed by the number of sessions completed on the WeChat mini program and the number of weekly nurse support sessions attended by participants.
Intervention acceptability | 6 weeks post-randomization
  The Intervention acceptability will be assessed via semi-structured qualitative interviews conducted with trial participants after the intervention.
Intervention fidelity | 6 weeks post-intervention
  Throughout the study, all nurse support sessions will be recorded. A random sample of 20% of the sessions will be evaluated by a psychologist for treatment fidelity using a modified version of the Yale Adherence and Competence Scale.

IPD SHARING:
Plan to Share IPD: Undecided